CLINICAL TRIAL: NCT05850286
Title: VRd-based Regimen Combined With CART-ASCT-CART2 as First-line Therapy for Newly Diagnosed Multiple Myeloma Patients With P53 Abnormalities：a Prospective, One-arm, Single-center Phase II Study
Brief Title: A Study of VRd-based Regimen Combined With CART-ASCT-CART2 Treatment in NDMM Patients With P53 Abnormalities
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022063（2）
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VRD-based Regimen Combined With CART-ASCT-CART2 (Experimental): Autologous BCMA-directed CAR-T cells, Double infusion intravenously at a target dose of 2-4 x 10^6 anti-BCMA CAR+T cells/kg respectively.
  Participants will receive VRD-based regimen induction, first CAR-T infusion, consolidation, ASCT and second CAR-T infusion. Maintenance therapy was initiated on day 100 and entered the follow-up period.
  Interventions: Biological: anti-BCMA CAR-T; Drug: VRD-based Regimen

INTERVENTIONS:
Biological: anti-BCMA CAR-T — Autologous BCMA-directed CAR-T cells, double infusion intravenously at a target dose of 2.0-4.0 x 10^6 anti-BCMA CAR+T cells/kg.
Drug: VRD-based Regimen — Bortezomib, Lenalidomide and Dexamethasone

SUMMARY:
This is a single-arm, open-label study to evaluate the efficacy and safety of VRD(Bortezomib, Lenalidomide and Dexamethasone)-based regimen combined with CART-ASCT-CART2 in patients with newly diagnosed multiple myeloma with p53 gene abnormalities.

DETAILED DESCRIPTION:
The study is a prospective, single-arm, single-centre, phase II study designed to evaluate the efficacy and safety of treatment with the VRd (short for Bortezomib, Lenalidomide, Dexamethasone)-based regimen in combination with the CART-ASCT-CART2 in newly diagnosed multiple myeloma patients with P53 gene abnormalities. Patients received 3 courses of induction therapy with VRd-based regimen followed by a first infusion of CAR-T cells. Patients then received 3 courses of consolidation therapy, followed by ASCT and second infusion of CAR-T cells. R maintenance therapy starts on day 100 after ASCT

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent (ICF) .
2. Age ≥ 18 years and ≤ 65 years.
3. Meet the internationally accepted Criteria for the diagnosis of newly diagnosed multiple myeloma (Chinese guidelines for the diagnosis and management of multiple myeloma (revised in 2022) criteria)
4. Patients have not received previous anti-multiple myeloma-related chemotherapy, have not received previous extensive pelvic radiotherapy (more than half of the pelvic area), and have not received previous anti-multiple myeloma hormone therapy, except for those who have used hormones for no more than 14 days for symptom control.
5. The patient have one or more measurable multiple myeloma lesion, must include one of the following conditions:

   * Serum M protein≥1.0 g/dL(10g/L)
   * Urine M protein≥200 mg/24h
   * Serum free light chain(sFLC): κ/λ FLC ratio is abnormal and affected FLC ≥10mg / dL
6. p53 gene abnormalities: Plasma cells were enriched by CD138 immunomagnetic and then detected by FISH. Cut-off ≥20%., or P53 mutation by second-generation sequencing.
7. ECOG scores 0 - 1;
8. No active infection
9. All screening blood biochemistry: tests should be performed according to the protocol and within 14 days before enrollment. Screening laboratory values must meet the following criteria： a.TBIL<1.5 x upper limit of normal (ULN) (<3 x ULN in patients with Gilbert's syndrome); b.AST and ALT <3 x ULN.; c. Creatinine clearance ≥ 60mL/min (calculated using Cockroft-Gault formula).
10. normal pulmonary function and oxygen saturation ≥ 92% on room air.
11. Routine blood tests (performed within 7 days, no RBC transfusion, no G-CSF/GM-CSF/platelet agonists, no drug correction within 14 days before screening, no PLT transfusion within 7 days) : WBC ≥ 1.5 x 109/L, ANC ≥ 1.0 x 109/L, Hb ≥ 85 g/L PLY ≥ 75 x 109/L (if BMPC < 50%) or PLT ≥ 50 x 109/L (if BMPC ≥ 50%)
12. Patients must be able to take prophylactic anticoagulant therapy as recommended by the study.
13. The woman is not breastfeeding, is not pregnant and agrees not to be pregnant during the study period and for the following 12 months. Male patients agreed that their spouse would not become pregnant during the study period and for 12 months thereafter.
14. Willing and able to complete the study procedures and follow-up examinations.

Exclusion Criteria:

1. Plasma cell leukemia.
2. Documented active amyloidosis.
3. Multiple myeloma with central nervous system (CNS) invasion
4. Unsuitable for autologous stem cell transplantation, such as severe cardiopulmonary disorders
5. Patients with peripheral neuropathy greater than grade 2 or peripheral neuropathy greater than grade 2 with pain at baseline, regardless of whether they were currently receiving medical therapy
6. Known intolerance, hypersensitivity, or contraindication to BCMA-CART cellular products.
7. Patients with unstable or active cardiovascular system disease, meeting any of the following:

   1. Unstable angina pectoris, symptomatic myocardial ischaemia, myocardial infarction or coronary artery reconstruction within 180 days prior to the first dose.
   2. Uncontrolled hypertension (>140/90 mmHg with blood pressure fluctuations of more than 180/100 mmHg over a 6-month period).
   3. Uncontrolled and clinically significant conduction abnormalities (e.g. patients with ventricular arrhythmias controlled by antiarrhythmic medication), not excluding patients with 1st degree atrioventricular (AV) block or asymptomatic left anterior bundle branch block/right bundle branch block (LAFB/RBBB)).
   4. Congestive heart failure (CHF) classification ≥ grade 3 as defined by the New York Heart Association (NYHA).
   5. Left ventricular ejection fraction (LVEF) <50% on echocardiography.
   6. History of stroke or intracranial haemorrhage within 12 months prior to screening.
   7. Presence of a serious thrombotic event prior to treatment.
8. Known positive serology for HIV or HIV seropositivity.
9. Active hepatitis B or C infection. Screening requires serologic testing for hepatitis. If hepatitis B surface antigen and hepatitis B core antibody were positive, a negative DNA polymerase chain reaction (PCR) result was needed before enrollment (after anti-hepatitis B therapy, a negative DNA polymerase PCR result was confirmed before enrollment). If the hepatitis C antibody was positive, the RNA PCR test should be negative prior to enrollment
10. Life expectancy of <3 months
11. Women who are pregnant or breastfeeding
12. Any active gastrointestinal dysfunction that affects the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that may affect the absorption of the studied treatment medication
13. Subjects had major surgery within 2 weeks before randomization (for example, general anesthesia), or is not fully recovered from the surgery, or surgery is arranged during study period.
14. Received live attenuated vaccine within 4 weeks prior to study treatment.
15. According to the researcher's judgement, any condition including but not limited to serious mental illness, medical illness or other symptoms/conditions that may affect study treatment, compliance, or the capability of providing informed consent.
16. Necessary medication or supportive therapy is contraindicated with study treatment.
17. Any diseases or complications that may interfere with the study.
18. Patients are not willing to or cannot comply with study scheme.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
complete response rate (CRR) | after induction therapy, 1 month after the first CAR-T cell transfusion, the consolidation therapy ends, 12 months after the second CAR-T cell transfusion
  CRR(including sCR / CR , based on IMWG 2016 efficacy evaluation criteria)
Overall response rate (ORR) | after induction therapy, 1 month after the first CAR-T cell transfusion, the consolidation therapy ends, 12 months after the second CAR-T cell transfusion
  ORR(including sCR / CR / VGPR / PR, based on IMWG 2016 efficacy evaluation criteria)
Negative MRD rate | after induction therapy, 1 month after the first CAR-T cell transfusion, the consolidation therapy ends, 12 months after the second CAR-T cell transfusion
  Rate of negative minimal residual disease
Overall Survival (OS) | 1 year
  Occurrence of death regardless of cause
Progression free survival (PFS) | 1 year
  Duration from start of study treatment to PD or death (regardless of cause), whichever comes first
Duration of Remission(DOR) | 2 year
  Duration from the first evaluation of at least partial remission (PR) to the onset of disease progression or death due to disease progression (whichever occurs first)

SECONDARY OUTCOMES:
The incidence of treatment-emergent adverse events (TEAEs) | 2 year
  The incidence of treatment-emergent adverse events (TEAEs)

OTHER OUTCOMES:
The CART cell duration in vivo | 1 year
  The copies of BCMA-CART DNA in peripheral blood with qPCR method

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China